CLINICAL TRIAL: NCT01838798
Title: Neuropsychological Impact of Hospitalization on Intubated, Ventilated and Sedated ICU Patients
Acronym: NeuroPsy Réa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LOCAL/2012/CR-02; 2013-A00022-43 (Other: RCB number)
Record Dates: First submitted 2013-04-21; First posted 2013-04-24 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2016-10

CONDITIONS: Stress Disorders, Post-Traumatic; Depression
Keywords: cognitive disorders; quality of life; Intensive care
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Cognitive Dysfunction | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study population (Experimental): See in inclusion/exclusion criteria.
  Interventions: Baseline activities; Clinical interview with a psychologist; Telephone interview 2 months after ICU discharge; Clinical interview with a psychologist .
  Interventions: Other: Baseline activities; Other: Clinical interview with a psychologist; Other: Telephone interview 2 months after ICU discharge

INTERVENTIONS:
Other: Baseline activities — Initial consent procedures and baseline data collection.
Other: Clinical interview with a psychologist — Clinical interview with a psychologist.
  This interview with a psychologist will take place after patient consent procedures, and at least 2 days after discontinuation of sedation, and before leaving the ICU. This interview will include:
  * An inventory of peritraumatic distress symptoms
  * A questionnaire on peritraumatic dissociative experiences
  * An assessment of related, potential impacts
  * The HADS questionnaire
Other: Telephone interview 2 months after ICU discharge — At 2 months after leaving the ICU, a psychologist will contact the patient with questions regarding his/her representation of hospitalization. This implies the following:
  * Questionnaires assessing memories and stressors (Questionnaires ICUMT, and ICU-SEQ
  * An assessment of psychological trauma
  * An assessment of potential impacts
Other: Clinical interview with a psychologist — At 4 months after ICU discharge, the patient has a clinical interview during which a psychologist will:
  * assess cognitive functions
  * evaluate clinical symptoms of depression
  * assess quality of life
  * assess symptoms of post traumatic stress

SUMMARY:
This is a prospective, single-center, pilot, cohort study. The first phase of this study is observational and the usual care of patients is maintained during the ICU stay, except for an interview with a psychologist preceding patient discharge. A phone interview at 2 months and a visit with a psychologist at four months after ICU discharge are specific to the study.

The main objective of this study is to make a first estimate of the percentage of patients (CI = +- 10%) with cognitive impairment at four months after ICU discharge. The presence / absence of cognitive impairment will be determined by the D2 test.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. To study the potential links between cognitive impairment and quality of life 4 months after discharge from the Intensive Care Unit.

B. To study the associations between variables measured during hospitalization. Is there "clustering" among certain symptoms during hospitalization?

C. To study the associations between variables measured at two and four months after ICU discharge. Is there clustering among these symptoms?

D. To study potential risk factors for cognitive problems at 4 months after ICU discharge.

E. If objective C determines the presence of clusters, is the presence / absence of these clusters related to the variables (or clusters of variables) measured during hospitalization?

F. To study potential risk factors for poor quality of life at 4 months:

ELIGIBILITY:
Inclusion Criteria:

* The patient (or his/her "trusted person") must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for a telephone interview at 2 months after ICU discharge, and for a follow-up visit at 4 months after ICU discharge
* Patient admitted to the ICU and intubated and ventilated for at least 48 hours

Exclusion Criteria:

* The patient is currently participating in or has participated in another study (within the past 3 months) that might influence the results of the current study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient has a contra-indication for a treatment used in this study
* Patient admitted to intensive care with sedation started for more than 24 hours
* Patient with neurological or psychiatric (cognitive) disorders
* Patient admitted for cardiac arrest
* Patient admitted for stroke
* Patient admitted for cervical trauma > C6
* Patient presenting with tracheotomy accompanied by long-term mechanical ventilation
* Moribund patient or with little hope of survival beyond 48 hours
* Patients for whom a limitation or termination of care is considered
* McCabe Score = 0
* Knauss Scale = C or D

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2013-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Presence/absence of cognitive impairment | 4 months after ICU discharge
  based on D2 test

SECONDARY OUTCOMES:
Duration of sedation | expected average of 48 hours
Duration of ventilation | expected average of 36 hours
Daily average for RASS scale | Expected maximum of 28 days
Daily average for Behaviour pain scale | expected average of 48 hours
CAM ICU score | upon awakening (expected average of 48 hours)
Peritraumatic distress inventory | expected average of 5 days (end of ICU stay)
Questionnaire PDEQ-10 | expected average of 5 days (end of ICU stay)
Assessment of potential impacts | expected average of 5 days (end of ICU stay)
HADS score | expected average of 5 days (end of ICU stay)
ICUMT questionnaire | 60 +- 3 days after ICU discharge
ICU-SEQ questionnaire | 60 +- 3 days after ICU discharge
Assessment of psychotramatisme | 60 +- 3 days after ICU discharge
HADS score | 60 +- 3 days after ICU discharge
PCLS scale (DSM IV items) | 4 months after ICU discharge
IDS-C Questionnaire | 4 months after ICU discharge
SF-36 | 4 months after ICU discharge
Forward span test | 4 months after ICU discharge
Backwards span test | 4 months after ICU discharge
Rey 15-word test | 4 months after ICU discharge
Test D2 (units = n) | 4 months after ICU discharge
Wisconsin test | 4 months after ICU discharge
Stroop test | 4 months after ICU discharge
Verbal fluency test | 4 months after ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Justine Pereira, Study Director — Centre Hospitalier Universitaire de Nîmes; Claire Roger, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France